CLINICAL TRIAL: NCT01615211
Title: A Randomized Pilot Study of Two New Drug Combinations Fot the Termination fo Early Pregnancy
Brief Title: Randomized Study of Letrozole and Trilostane for Medical Abortion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No access to study drug Trilostan. Company closed down
Sponsor: Kristina Gemzell Danielsson (Other)
Collaborators: Karolinska Institutet (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W300TL
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Medical Abortion, Complete or Unspecified, Without Complication
Keywords: Abortion; medical abortion; termination of pregnancy; Mifepristone; misoprostol; letrozole; trilostane; femara; Modrenal
MeSH Terms: interventions — Letrozole; trilostane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard treatment (No Intervention): patients will receive standard treatment with 200mg Mifepristone and after 36-48 hours 800 mcg of misoprostol vaginally
- trilostane (Active Comparator): patients will receive Day 1: Mifepristone 200 mg and Trilostane 120mg 1 tablet twice and Day 2 Trilostane 240mg twice. On Day 3 800 mcg misoprostol will be given vaginally.
  Interventions: Drug: Trilostane
- Letrozole (Active Comparator): Patients will receive on Day 1 Mifepristone 200mg and Letrozole 2,5mg 3 tablets and on Day 2 Letrozole 2,5mg 3 tablets. On day 3 800mcg of misoprostol will be given vaginally
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Day 1 Letrozole 2,5mg 3 tablets Day 2 Letrozole 2,5mg 3 tablets
  Other Names: Brand name Femar
  Arms: Letrozole
Drug: Trilostane — Day 1 Trilostane 120mg twice and Day 2 Trilostane 240mg twice
  Other Names: Brand name Modrenal
  Arms: trilostane

SUMMARY:
In menstruation an effective shedding of the endometrial lining occurs. Both progesterone and estrogen levels fall sharply at this time. During medical abortion the endometrial shedding is sometimes ineffective causing an incomplete abortion which may cause prolonged bleeding or require surgical intervention. In medical abortion a progesterone antagonist is used as treatment but the estrogen levels are not targeted. The investigators wish to explore whether addition of letrozole or trilostane which target estrogen levels can lead to a more effective shedding of the endometrial lining.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-45 without any contraindication for treatment of any of the drugs involved in teh study

Exclusion Criteria:

* Any ongoing medication or medical condition smoking >20 cigarettes per day BMI >30

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
efficacy | 4 weeks
  Evaluation of complete abortion by clinical judgement and ultrasonography

SECONDARY OUTCOMES:
Acceptability | 1 week, 2 weeks and 4 weeks
  questionnaire. Preferred future method of medical abortion.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, professor, Principal Investigator — Karolinska Institutet; Helena Kopp Kallner, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden